CLINICAL TRIAL: NCT01226589
Title: The Impact of Pharmacist Discharge Medication Reconciliation on Unintentional Medication Discrepancies From Inpatient Discharges at the Alberta Cancer Board Cross Cancer Institute
Brief Title: Pharmacist Discharge Medication Reconciliation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Health services (Other)
Responsible Party: Carole Chambers, Alberta Cancer Board
Organization: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23851
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Medication Reconciliation
Keywords: Cancer cancer; MRS; Treatment response; Histologically confirmed diagnosed Breast cancer.; Patient is 18 years or older.; Karnofsky performance score is equal to or greater than 70.; No previously irradiated or recurrent breast.; No contraindication to MRS/MRI.
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: MRS

SUMMARY:
Adverse drug events can occur commonly due to medication errors during the transition of care in a health care facility. Medication reconciliation is the process of comparing medications and providing an accurate medication list as a resource for prescribers, which is currently only being done upon inpatient admission at the CCI. The purpose of this study is to see if pharmacist medication reconciliation at discharge reduces unintentional medication discrepancies for inpatient discharges.

ELIGIBILITY:
Inclusion Criteria:

* Cancer inpatients under the care of Dr. Follett or Dr. Candler
* Cancer inpatients to be discharged from the CCI
* Patients >18 years of age
* Patients that are taking >1 medications or herbals total at home.

Exclusion Criteria:

* Cancer inpatients that are considered radioactive or in "hot rooms" (ie. Selectron patients or patients receiving radiation treatment for thyroid)
* Patients that do not remain in hospital >72 hours
* Patients without a home phone number or equivalent contact number.
* Language barrier (patients unable to speak or understand English).
* Patients that are readmitted and already included into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
MRS Correlation with Treatment Response. | up to 1 year
  The percentage of patients with at least one unintentional medication discrepancy after discharge from the Cross Cancer Institute

SECONDARY OUTCOMES:
Correlation with Tumor Stage | up to 1 year
  The amount of medication discrepancies after discharge that has the potential to cause moderate harm to severe harm.
The frequency of each type of unintentional medication discrepancies.

CONTACTS AND LOCATIONS:
Overall Officials: Carole Chambers, BSc. Pharmacy, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada